CLINICAL TRIAL: NCT03156712
Title: Serum Iron Increase With From Iron-enriched Aspergillus Compared to Ferrous Sulfate in Healthy Female Subjects
Brief Title: Iron Absorption From Iron-enriched Aspergillus Oryzae
Acronym: BIEFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIEFS
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Iron-deficiency; Absorption; Iron; Anemia, Iron Deficiency; Bioavailability; Serum Iron
Keywords: Anemia; Iron deficiency anemia; Iron fortification; ferrous sulfate; aspergillus oryzae; iron supplementation; AUC
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferrous sulfate; aspartyl-aspartic acid

STUDY DESIGN:
Intervention Model Description: Double-blinded, cross-over experimental design, whereby subjects were randomly given three different iron supplements with a meal in three different visits. All three visits (iron treatments) were each separated by two weeks time.
Who Masked: Participant, Investigator
Masking Description: Both investigators and participants were blinded to the iron treatment in this double-blinded, crossover study. Three different iron supplements were given, whereby participants were either administered 10 mg FeSO4, 10 mg ASP Fe, or 20 mg ASP Fe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FeSO4 (Experimental): Ferrou sulfate: Each participant was given a one time oral dose of the 10 mg iron as ferrous sulfate with the test meal (described in study design) and serum iron was measured every 30 min for 4 hours.
  Interventions: Dietary Supplement: Ferrous sulfate
- ASP Fe (10 mg) (Experimental): ASP (10 mg Fe): Each participants was given a one time oral dose of ASP containing 10 mg iron. The capsule was consumed with the test meal and serum iron was measured every 30 min for 4 hours.
  Interventions: Dietary Supplement: Ferrous sulfate
- ASP Fe (20 mg) (Experimental): ASP (20 mg Fe): Each participant was given a one time oral dose ASP containing of 20 mg iron The capsule was consumed with the test meal and serum iron was measured every 30 min for 4 hours.
  Interventions: Dietary Supplement: Ferrous sulfate

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — The intervention is the ASP, a natural form of iron supplement and compared to a widely used dietary iron supplement ferrous sulfate in terms of serum iron response over a 4h period.
  Other Names: ASP (10 mg); ASP (20 mg)

SUMMARY:
Ferrous sulfate is rapidly absorbed and the bolus of iron enters blood rather quickly possibly leading to higher concentrations of non-transferrin bound iron which induces oxidative stress. The objective of this study was to determine how quickly iron enters into blood stream from the iron-enriched Asperigillus oryzae (AspironTM, ASP) in contrast to ferrous sulfate. Seventeen healthy, female subjects (18-35 y) were randomized, double blind, cross-over experimental design with three treatments: 10 mg iron as FeSO4 and ASP as well as 20 mg iron as ASP.

DETAILED DESCRIPTION:
In a double-blinded cross-over design, 17 research participants were randomly given one of three iron-treatments : ferrous sulfate (10mg), AspironTM (10mg), and AspironTM (20mg). Each iron treatment was given with a test meal consisting of cabbage, green peas, green beans, soy sauce, peanut oil, 40 g baby carrots, steamed rice, and orange juice. Each subject consumed a meal with one of the three iron supplements in a random order and all participants consumed the three supplements 2 weeks in between each treatment. Prior to consuming the test meal with iron supplement for each treatment, blood was collected for baseline serum iron measuremt. Following consumption of the meal with iron, subsequent blood draws were taken every 30 minutes over the time period of 4 hours to assess the incease in serum iron. Ferritin, hepcidin, iron , and c-reactive protein concentrations were measured in the serum at baselime. After two weeks other treatments were administered to each participant. The serum iron response curves for each treatment were constructed and the area under the curve (AUC) was calculated with the change of serum iron from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* Non-lactating
* Non-smoker
* Not taking medications
* Not taking dietary supplements (vitamins or minerals)
* No history of gastrointestinal conditions

Exclusion Criteria:

* Any history of gastrointestinal conditions
* On medications that interfere with iron absorption
* Unwilling to stop taking dietary supplements (vitamins or minerals)
* Pregnant
* Lactating
* Smoker

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2013-11-20 (Actual); Study Completion 2014-02-13 (Actual)

PRIMARY OUTCOMES:
Serum iron | 12 hours
  Area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Manju B Reddy, Ph.D., Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Publish a paper